CLINICAL TRIAL: NCT00713479
Title: A Human Laboratory Assessment of the Safety and Potential Efficacy of Varenicline in Methamphetamine-dependent Volunteers Receiving Methamphetamine
Brief Title: An Assessment of the Safety of Varenicline in Methamphetamine-dependent Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steve Shoptaw, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18185-PI-EDL-V; P50DA018185 (NIH); DPMC (Other: NIH / NIDA)
Record Dates: First submitted 2008-07-10; First posted 2008-07-11 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Methamphetamine Addiction; Crystal Meth Addiction; Amphetamine Addiction
Keywords: methamphetamine; varenicline; Chantix; stimulant; crystal meth
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Sugar pill (placebo) drug dosing will begin at 0.5 mg once daily for the first 3 days of condition and will be increased to 0.5 mg twice daily for days 5-6 of this condition, and increased to 1 mg twice daily on days 7-10 of this condition.
  Interventions: Drug: Varenicline, then placebo; Drug: Placebo, then varenicline
- Varenicline (Active Comparator): Varenicline dosing will begin at 0.5 mg once daily for the first 3 days of condition and will be increased to 0.5 mg twice daily for days 5-6 of this condition, and increased to 1 mg twice daily on days 7-10 of this condition.
  Interventions: Drug: Varenicline, then placebo; Drug: Placebo, then varenicline

INTERVENTIONS:
Drug: Varenicline, then placebo — Subjects receive MA infusions on certain days first under varenicline (10 days) then under placebo (8 days) after a 14-24 day washout in order to determine study medication safety and tolerability
  Other Names: varenicline
Drug: Placebo, then varenicline — Subjects receive MA infusions on certain days first under placebo (10 days) then under varenicline(8 days) after a 14-28 day washout in order to determine study medication safety and tolerability
  Other Names: placebo

SUMMARY:
More people worldwide use amphetamine-type stimulants than any illicit drug besides cannabis, and methamphetamine (MA) abuse and dependence is the fastest growing drug problem in the United States. Much work remains in identifying an effective pharmacotherapy for MA dependence. The neurobiological actions produced by MA involve dopamine (DA), serotonin, and norepinephrine, but also include alterations to cholinergic neurotransmitter systems. Candidate compounds that target acetylcholine (ACh) are attractive options for development that have not received adequate attention. Varenicline is a drug that increases the release of DA in the brain and it is logical to assume that it would to some extent compensate for the reduction in these neurotransmitters that occurs in MA withdrawal.

Current research has linked certain genes that are related to neurotransmitters with drug abuse and memory impairment (e.g., A1 allele for the D2 dopamine receptor and catechol-O-methyltransferase). We will take blood samples and test for these genes in order to relate the findings to brain function.

This is a double-blind, placebo-controlled, within-subjects study to determine the safety and tolerability of MA in MA-dependent volunteers treated with varenicline and placebo.

DETAILED DESCRIPTION:
Study Procedures:

Study participants are those who meet criteria for MA dependence, who are not seeking treatment, and who also meet criteria for nicotine dependence. Participants will be asked to wear a telemetry device during screening and throughout the study that records heart rate and body temperature. Participants will be required to refrain from smoking at certain times, illicit and prescription drug use for the duration of the study and this will be confirmed with daily urine testing.

The study consists of 30 days or less of outpatient screening. The 2-component inpatient portion of the study lasts a total of 18 days. Participants will be admitted to the GCRC at UCLA for Days 1-10. After the first study day, participants will be randomized to varenicline or matched placebo for 9-days and then discharged from the GCRC. Then, after 2-4 weeks, the same subjects return to the GCRC to be switched to the alternate condition (placebo or varenicline) for the second component of the study, which lasts another 8-days. Each subject is randomized to both varenicline and placebo, so total time commitment is 18 inpatient study days. One follow-up visit is scheduled 2 weeks after completion of both study phases for assessment of delayed adverse events and for final payment.

On the first day of the inpatient procedure, subjects received 10 3mg infusions of methamphetamine over 2.5 hours for assessment of drug tolerability. On day 9 of the first component and day 7 of the second component, subjects received either 10 3mg infusions of saline OR methamphetamine over 2.5 hours. In the afternoon, the infusion was the opposite of the morning condition.

ELIGIBILITY:
Inclusion Criteria:

1. Be English-speaking volunteers who are not seeking treatment at the time of the study;
2. Be between 18-55 years of age;
3. Meet DSM-IV TR criteria for MA dependence;
4. Must be cigarette smokers, defined as smoking 10 or more cigarettes per day by self-report;
5. Have a self-reported history of using MA by the smoked or IV route and provide at least one MA-positive urine prior to admission;
6. Have vital signs as follows: resting pulse between 50 and 90 bpm, blood pressures between 105-150 mm Hg systolic and 45-90 mm Hg diastolic; this criterion must be met within 2 days of admission;
7. Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) < 2 x the upper limit of normal;
8. Have a baseline EKG that demonstrates normal sinus rhythm, normal conduction (including QTc), and no clinically significant arrhythmias;
9. Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician or nurse practitioner and the principal investigator.

Exclusion Criteria:

1. Have any history or evidence suggestive of seizure disorder or brain injury
2. Have any previous medically adverse reaction to MA, including loss of consciousness, chest pain, or epileptic seizure
3. Have neurological or psychiatric disorders, such as

   * psychosis, bipolar illness or major depression as assessed by SCID;
   * organic brain disease or dementia assessed by clinical interview;
   * history of any psychiatric disorder which would require ongoing treatment or which would make study compliance difficult;
   * history of suicide attempts within the past three months assessed by SCID and/or current suicidal ideation/plan as assessed by SCID;
4. Have evidence of clinically significant heart disease or hypertension, as determined by the PI;
5. Have a family history in first-degree relatives of early cardiovascular morbidity or mortality, as determined by the PI;
6. Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease;
7. Have HIV and are currently symptomatic, have a diagnosis of AIDS, or are receiving antiretroviral medication;
8. Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, upon hospital admission, and at the end of study participation;
9. Have asthma or currently use alpha or beta agonists, theophylline, or other sympathomimetics;
10. Have any other illness, condition, or use of psychotropic medications, which in the opinion of the PI and/or the admitting physician or nurse practitioner would preclude safe and/or successful completion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edythe D London, PhD, Principal Investigator — UCLA NPI
Locations (1):
- UCLA NPI, Los Angeles, California, United States

REFERENCES:
- [Result] Zorick T, Sevak RJ, Miotto K, Shoptaw S, Swanson AN, Clement C, De La Garza R 2nd, Newton TF, London ED. Pilot safety evaluation of varenicline for the treatment of methamphetamine dependence. J Exp Pharmacol. 2009 Dec 24;2:13-8. eCollection 2010. PMID 27186086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject were recruited from local advertisements for non-treatment seeking methamphetamine users in 2008.
Pre-assignment Details: Participants had 30 days in which to complete all eligibility procedures. Volunteers were: MA dependent who were not seeking treatment;nicotine dependent (smoking 10+ cigarettes/day);reported using MA via smoking or IV;could not have significant medical illnesses;be taking psychotropic medications or dependence criteria for other substances.
Groups:
- Placebo, Then Varenicline: Placebo drug dosing will begin at 0.5 mg once daily for the first 3 days of condition and will be increased to 0.5 mg twice daily for days 5-6 of this condition, and increased to 1 mg twice daily on days 7-10 of this condition. After a 14-28 day washout, the varenicline condition is started. Varenicline is taken daily for 10 days in the presence of 30 mg IV methamphetamine and 30 mg IV saline (infusion blinded to both study participants and staff members).
- Varenicline, Then Placebo: Varenicline dosing will begin at 0.5 mg once daily for the first 3 days of condition and will be increased to 0.5 mg twice daily for days 5-6 of this condition, and increased to 1 mg twice daily on days 7-10 of this condition. After a 14-28 day washout, the placebo condition is started. Placebo is taken daily for 10 days in the presence of 30 mg IV methamphetamine and 30 mg IV saline (infusion blinded to both study participants and staff members).
Period: First Medication Condition
Arm/Group | Placebo, Then Varenicline | Varenicline, Then Placebo
Started | 6 | 6
Completed | 2 | 6
Not Completed | 4 | 0
Period: Washout
Arm/Group | Placebo, Then Varenicline | Varenicline, Then Placebo
Started | 2 | 6
Completed | 2 | 6
Not Completed | 0 | 0
Period: Next Medication Condition
Arm/Group | Placebo, Then Varenicline | Varenicline, Then Placebo
Started | 2 | 6
Completed | 2 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a crossover design wherein each subject completed both the sugar pill treatment condition and the varenicline(medication under study) condition. Two subjects in the placebo condition did not complete the first component of the trial.
Groups:
- Total Sample: Includes only subjects who completed both components of the trial.
Arm/Group | Total Sample
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — This value is for subjects completing both arms of the trial (n=8)
  years | 39.3 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure is evaluated at 15 min intervals under placebo or varenicline in the presence of methamphetamine over 140 minutes post infusion. Data is pooled and the mean and standard deviation are presented.
Time Frame: 15 minute intervals
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: time points
Groups:
- Sugar Pill: Study drug dosing will begin at 0.5 mg once daily for the first 3 days of condition and will be increased to 0.5 mg twice daily for days 5-6 of this condition, and increased to 1 mg twice daily on days 7-10 of this condition.
  Sugar pill : Medication is taken daily for 10 days in the presence of 30 mg IV methamphetamine and 30 mg IV saline (infusion blinded to both study participants and staff members).
- Varenicline: Study drug dosing will begin at 0.5 mg once daily for the first 3 days of condition and will be increased to 0.5 mg twice daily for days 5-6 of this condition, and increased to 1 mg twice daily on days 7-10 of this condition.
  Varenicline : Medication is taken daily for 10 days in the presence of 30 mg IV methamphetamine and 30 mg IV saline (infusion blinded to both study participants and staff members)
Arm/Group | Sugar Pill | Varenicline
Number analyzed (Participants) | 8 | 8
Number analyzed (time points) | 80 | 80
mm Hg | 126.4 (12.1) | 127.4 (8)

2. Primary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure is evaluated at 15 min intervals under placebo or varenicline in the presence of methamphetamine over 140 minutes post infusion. Data is pooled and the mean and standard deviation are presented.
Time Frame: 15 minute intervals
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: Time Points
Groups:
- Sugar Pill; Varenicline: Study drug dosing will begin at 0.5 mg once daily for the first 3 days of condition and will be increased to 0.5 mg twice daily for days 5-6 of this condition, and increased to 1 mg twice daily on days 7-10 of this condition.
  Medication is taken daily for 10 days in the presence of 30 mg IV methamphetamine and 30 mg IV saline (infusion blinded to both study participants and staff members).
Arm/Group | Sugar Pill | Varenicline
Number analyzed (Participants) | 8 | 8
Number analyzed (Time Points) | 80 | 80
mm Hg | 72.4 (6.6) | 71.7 (4.3)

3. Primary Outcome: Heart Rate
Description: Heart rate is evaluated at 15 min intervals under placebo or varenicline in the presence of methamphetamine over 140 minutes post infusion. Data is pooled and the mean and standard deviation are presented.
Time Frame: 15 minute intervals
Measure: Mean (Standard Deviation); unit: bpm
Units Other Than Participants: Time Points
Arm/Group | Sugar Pill | Varenicline
Number analyzed (Participants) | 8 | 8
Number analyzed (Time Points) | 80 | 80
bpm | 80.4 (8.8) | 84.4 (9.3)

4. Secondary Outcome: Depression
Description: Using the Beck Depression Index (BDI-II), depression was assessed on a daily basis. The daily mean score during the medication intervention period is presented, with a lower score indicating lower reported depression. The scores range from 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; and 29-63: severe depression.
Time Frame: Daily
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Total BDI
Arm/Group | Sugar Pill | Varenicline
Number analyzed (Participants) | 8 | 8
Number analyzed (Total BDI) | 64 | 64
units on a scale | 2.3 (2.5) | 2.5 (3.3)

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Varenicline
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/8 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=8) | Varenicline (N=8)
Insomnia (Nervous system disorders) | 4 (4) | 6 (6)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Asymptomatic PVCs (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu-like Symptoms (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Depressed Mood (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes